CLINICAL TRIAL: NCT07302269
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics of a Single Oral Dose of VV261 Tablets in Chinese Healthy Volunteers
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics of VV261 Tablets in Chinese Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VV261-01
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: VV261; Phase I; Tolerability; Pharmacokinetic; Safety
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VV261 (Experimental)
  Interventions: Drug: VV261 5mg group; Drug: VV261 20mg Group; Drug: VV261 50mg group; Drug: VV261 100mg group; Drug: VV261 150mg group; Drug: VV261 300mg group; Drug: VV261 500mg group; Drug: VV261 750mg group; Drug: VV261 1000mg group
- Placebo (Placebo Comparator)
  Interventions: Drug: VV261 20mg Group; Drug: VV261 50mg group; Drug: VV261 100mg group; Drug: VV261 150mg group; Drug: VV261 300mg group; Drug: VV261 500mg group; Drug: VV261 750mg group; Drug: VV261 1000mg group

INTERVENTIONS:
Drug: VV261 5mg group — 2 subjects will receive VV261 5mg, orally
  Arms: VV261
Drug: VV261 20mg Group — 6 subjects receive VV261 20mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 50mg group — 6 subjects receive VV261 50mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 100mg group — 6 subjects receive VV261 100mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 150mg group — 6 subjects receive VV261 150mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 300mg group — 6 subjects receive VV261 300mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 500mg group — 6 subjects receive VV261 500mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 750mg group — 6 subjects receive VV261 750mg,orally; 2 subjects will receive placebo,orally.
Drug: VV261 1000mg group — 6 subjects receive VV261 1000mg,orally; 2 subjects will receive placebo,orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending-dose study to evaluate the safety, tolerability and pharmacokinetics characteristics of VV261 tablets in healthy adults.

DETAILED DESCRIPTION:
The study is designed to enroll 58 volunteers. The pilot study is an open-labelled study where both volunteers receive 5 mg VV261 tablets. The formal study, conducted as a double-blind study, comprise 7dose groups with 8 volunteers (both sexes) each. Volunteers will be randomly assigned to receive either the VV261 tablets or placebo in a ratio of 6:2. The formal study's dose groups are designed as 20 mg, 50 mg, 150 mg, 300 mg, 500 mg, 750 mg, and 1000 mg. Based on observed tolerability and safety data or obtained pharmacokinetic data, adjustments are allowed at all dose levels in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old, males or females;
2. Males weight no less than 50 kg, females weight no less than 45 kg, with body mass index of 19 to 26 kg/m^2;
3. Vital signs examination, physical examination, laboratory examination ,electrocardiogram examination chest CT and B-ultrasound of liver, gallbladder, pancreas, spleen, kidney and thyroid results are normal or considered abnormal without clinical significance by the investigator;
4. Volunteers who are willing to take proper contraceptive methods during the study and within 3 months after the the last administration;
5. Volunteers who are able to understand and follow the study protocol and instructions; volunteers who have voluntarily decided to participate in this study, and sign the informed consent form.

Exclusion Criteria:

1. Volunteers with hypersensitivity to preparation or any of the excipients;
2. Volunteers with allergic constitution (such as asthma, urticaria, eczematous dermatitis and other allergic diseases), or have a history of drug or food allergy;
3. Volunteers with central nervous system, cardiovascular system, gastrointestinal, respiratory system, urinary, hematologic, or metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;Volunteers with a history of gastrointestinal conditions that may impair drug absorption (e.g., gastrectomy or small intestine resection, atrophic gastritis, gastrointestinal ulcers or perforations/fistulas, gastrointestinal bleeding, or obstruction);
4. Volunteers with a history of diseases affecting bone marrow hematopoietic function or reducing immunological function (including leukemia, myelodysplastic syndrome, aplastic anemia, systemic lupus erythematosus, rheumatoid arthritis, etc.) or treatment history (tumor chemotherapy or radiotherapy, use of immunosuppressants, etc.);
5. Volunteers with a history of spleen diseases;
6. If any of the following parameters were considered abnormal with clinical significance: white blood cell count, red blood cell count, platelet count, reticulocyte count, and absolute neutrophil count;
7. If any of the following parameters were considered abnormal with clinical significance: total bilirubin, alkaline phosphatase, alanine aminotransferase, and aspartate aminotransferase;
8. Volunteers who have received blood transfusion or used blood products within 3 months before screening or who have lost more than ≥400 mL of blood due to other reasons (excluding menstruation);
9. Volunteers who have participated in clinical trials and received drugs within 3 months before screening;
10. Volunteers who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 2 weeks before screening;
11. Volunteers who have received vaccination within the first 2 weeks before screening, or planned to receive any vaccine during the trial or within 1 week after the end of the study;
12. Volunteers with a history of drug abuse within 1 year before screening or positive urine drug screening within 1 year before screening results (morphine, tetrahydrocannabinol, methamphetamine, dimethylene diphenazine , ketamine, and cocaine);
13. Volunteers who drink more than 14 standard units or at least twice a day per week within one year before screening,(one standard unit equals 200 mL of beer with 5% alcohol or 25 mL of white wine with 40% alcohol content or 85 mL of red wine with 12% alcohol);
14. Volunteers who smok more than 5 cigarettes a day within one year before screening;
15. Volunteers who can't quit smoking or drinking during the trial period;
16. Volunteers who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, treponema pallidum antibody or human immunodeficiency virus antibody (Anti-HIV);
17. Volunteers who cannot tolerate blood collection with intravenous indwelling needles or blood fainting;
18. Volunteers with lactose intolerance or cannot comply with a uniform diet (such as special dietary requirements, intolerance of standard meals, etc.), volunteers who have consumed excessive amounts of strong tea, coffee or caffeinated beverages in the 3 months before screening;
19. Volunteers with difficulty in swallowing tablets;
20. Pregnant or lactating women or male volunteers whose female partners plan to conceive within 3 months;
21. The investigator believes that there are other unsuitable factors to participate this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | 48 hours after administration]
  maximum observed plasma concentration
AUC0-t | 48 hours after administration
  area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | 48 hours after administration]
  area under the plasma concentration-time curve from time zero to infinity
Tmax | 48 hours after administration
  time at which Cmax occurs
t1/2 | 48 hours after administration
  half life of elimination
Kel | 48 hours after administration
  elimination rate constant
CLz/F | 48 hours after administration
  apparent clearance
Vd/F | 48 hours after administration
  apparent volume of distribution during the terminal phase
MRT | 48 hours after administration
  mean residence time
AE & SAE | from day1 to day7 after administration
  Adverse event & serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Anhui Medical University

IPD SHARING:
Plan to Share IPD: No